CLINICAL TRIAL: NCT03624322
Title: Phase1 Randomized, Double-Blind, Placebo/Active-Controlled, SAD, 2-Way, Incomplete Block, 2-Period Crossover, Safety, Tolerability, PK/PD Study of 3 Doses INP105 (Olanzapine Delivered by I231 POD® Device) Nasal Spray in Healthy Volunteers
Brief Title: Safety and Tolerability of INP105 (Olanzapine by I231 POD® Device) Nasal Spray in Healthy Volunteers - SNAP 101
Acronym: SNAP101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INP105-101
Record Dates: First submitted 2018-07-25; First posted 2018-08-10 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-08

CONDITIONS: Acute Agitation
Keywords: Agitation; Schizophrenia; Bipolar I disorder; OLZ; Olanzapine; Zyprexa; POD® device
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Intervention Model Description: Period 1 (n=36) assignment to 1 of 2 reference therapy treatment groups over 3 cohorts Period 2 (n=36) assignment to 1 of 3 IP treatment groups over 3 cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Period 1 (Active Comparator): Period 1 (n=36) assignment to 1 of 2 reference therapy treatment groups (Zyprexa 5mg IM or Zydis 10mg orally disintegrating wafer, 10mg) over 3 cohorts (single dose)
  Interventions: Drug: Zyprexa IM; Drug: Zydis
- Period 2 (Experimental): Period 2 (n=36) assignment to 1 of 3 IP treatment groups (INP105 of 5, 10, or 20mg or placebo) administered with the I231 POD® Device) over 3 cohorts (single dose)
  Interventions: Drug: INP105; Device: I231 POD® Device

INTERVENTIONS:
Drug: Zyprexa IM — 5mg
  Arms: Period 1
Drug: Zydis — 10mg orally disintegrating wafer
  Other Names: Zyprexa Zydis
  Arms: Period 1
Drug: INP105 — Single, ascending doses of 5, 10, or 20mg capsules OLZ (olanzapine) or placebo (MCC)
  Other Names: OLZ or placebo
  Arms: Period 2
Device: I231 POD® Device — Precision Olfactory Delivery (POD) device
  Other Names: POD®
  Arms: Period 2

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of INP105, which is an investigational drug-device combination product comprised of the drug component OLZ administered by a Precision Olfactory Delivery (POD®) nasal spray device (I231 POD® Device). The proposed indication for INP105 is the treatment of acute agitation associated with schizophrenia and bipolar I disorder.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo- and active-controlled, ascending-dose, 2-way, 2- period, incomplete block, crossover, Phase 1 trial to compare the safety, tolerability, PK and PD of 3 single doses of INP105 with the safety, tolerability, PK and PD of 1 dose of Zyprexa IM (5 mg) and 1 dose of oral Zyprexa Zydis (10 mg). Randomization for Periods 1 and 2 will occur for each subject on Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male (N=at least 9) and female (N=at least 9) 18 to 55 years of age (inclusive) at Screening, in good general health, with no significant medical history and no clinically significant abnormalities on physical examination at Screening or before first dose of IP.
2. Subjects must have a Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive.
3. Negative urine drug screen/alcohol breath test at Screening and Day -1. Repeat tests may be performed if false positive results are suspected.
4. Subjects must have the ability and willingness to attend the necessary visits at the study centre.
5. Written informed consent signed prior to entry into the study.
6. Female subjects of childbearing potential, and male subjects and their partners, must agree to use adequate contraception, defined as complete abstinence, documented evidence of surgical sterilization or condom plus approved contraceptive method

Exclusion Criteria:

1. Known hypersensitivity to Zyprexa IM, Zyprexa Zydis or any of the ingredients in them or in INP105 or the placebo.
2. Recently (within 3 months) or currently taking Zyprexa (any formulation).
3. Subjects taking medications known to inhibit or induce CYP1A2 at any time during the study period, and any subjects taking prescription medications, over the counter medications or supplements that, in the opinion of the Investigator, may impact the subject's response to INP105 or impact the subject's participation in the study. Oral contraceptives are permitted.
4. Subjects with medical history of hypotension or currently taking anti-hypertensives at Screening or throughout the study.
5. Current or recent smokers (<3 months since quitting); inadvertent one-off smokers and social smokers will also be excluded.
6. Females who are pregnant or lactating.
7. Subjects with any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the subject will comply with the study.
8. Abnormal and clinically significant laboratory test results.
9. History or presence of alcohol or drug abuse within the 2 years prior to the first IP administration.
10. Blood donation or significant blood loss within 60 days prior to the first IP administration.
11. Plasma donation within 7 days prior to the first IP administration.
12. Administration of IP in another trial within 30 days or 5 half-lives (whichever is longer) prior to the first IP administration.
13. Significant surgery within the past 3 months prior to the first IP administration determined by the Investigator to be clinically relevant.
14. Failure to satisfy the Investigator of fitness to participate for any other reason.
15. Acute illness within 30 days prior to Day 1. Subjects with minor viral illnesses (for example, upper respiratory tract infection) within 30 days prior to Day 1 may be randomized if all symptoms are resolved by admission and at the discretion of the Investigator.
16. Any nasal congestion, deviated septum, or physical blockage in either nostril.
17. Positive for human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult male (N=at least 9) and female (N=at least 9) 18 to 55 years of age (inclusive) at Screening
Enrollment: 38 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 30 days
  AEs and SAEs as assessed from baseline by physical exam, ECG, vital signs, and clinical laboratory results
PK profile of OLZ INP105 Tmax | 72 hours
  Tmax
PK profile of OLZ INP105 Cmax | 72 hours
  Cmax
PK profile of Zyprexa IM Tmax | 72 hours
  Tmax
PK profile of Zyprexa IM Cmax | 72 hrs
  Cmax
PK profile of Zyprexa Zydis Tmax | 72 hours
  Tmax
PK profile of Zyprexa Zydis Cmax | 72 hours
  Cmax
PD effects of INP105 vs placebo | 72 hours
  Changes in motor function measured by PD assessment compared to overall PK profile following ascending doses of INP105
PD effects of Zyprexa IM | 72 hours
  Changes in motor function measured by PD assessment compared to overall PK profile following a single dose of 5mg of Zyprexa IM
PD effects of Zyprexa Zydis | 72 hours
  Changes in motor function measured by PD assessment compared to overall PK profile following a single 10mg dose of Zyprexa Zydis oral disintegrating wafer

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Shrewsbury, MD, Study Director — Impel NeuroPharma; Niquita Tugiono, MD, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Shrewsbury SB, Hocevar-Trnka J, Satterly KH, Craig KL, Lickliter JD, Hoekman J. The SNAP 101 Double-Blind, Placebo/Active-Controlled, Safety, Pharmacokinetic, and Pharmacodynamic Study of INP105 (Nasal Olanzapine) in Healthy Adults. J Clin Psychiatry. 2020 Jun 30;81(4):19m13086. doi: 10.4088/JCP.19m13086. PMID 32609960